CLINICAL TRIAL: NCT05178784
Title: EEG Biomarker Study for Participants in the Neurolief "MOOD" Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Butler Hospital (Other)
Collaborators: Neurolief Ltd. (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 1823167
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active Stimulation: Adults exposed to active external Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) stimulation during the 8-week blinded treatment phase of the MOOD Clinical Trial (NCT04279522) who enrolled in this EEG substudy
  Interventions: Device: External Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) stimulation
- Sham Stimulation: Adults exposed to sham external Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) stimulation during the 8-week blinded treatment phase of the MOOD Clinical Trial (NCT04279522) who enrolled in this EEG substudy

INTERVENTIONS:
Device: External Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) stimulation — Relivion®DP is a device by Neurolief that delivers external, combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS), which is proposed as a novel treatment approach for MDD. The Relivion®DP device is designed for at-home self-administration by patients; it is comprised of a headset that holds electrodes, and it is worn externally on a person's head. When activated, the device delivers mild electrical stimulation pulses which can be managed by the user. The stimulation is intended to reduce MDD symptoms.
  Other Names: eCOT-NS
  Groups: Active Stimulation

SUMMARY:
This study will collect EEG data at 3 time points from up to 40 adults who are enrolled in a double clinical trial investigating a device that delivers noninvasive, self-administered external Combined Occipital and Trigeminal Neurostimulation (eCOT-NS) treatment for Major Depressive Disorder (Relivion®DP). Baseline (Pre-treatment) Frontal EEG Alpha Oscillations (Power) will be compared post-stimulation power.

DETAILED DESCRIPTION:
EEG Biomarkers may be useful for understanding abnormal brain oscillations associated with Major Depressive Disorder (MDD) and other psychiatric disorders as well as the brain changes that occur when symptoms remit. This study will invite adults with MDD who enroll and are randomized in the Neurolief Sponsored "MOOD" study to undergo collection of EEG data at pre-treatment baseline, again after completing the 8-week blinded treatment phase, and, if eligible/appropriate, again after completing an 8-week open-label treatment phase. EEG will be recorded at rest and during a computer task. This EEG "add-on" study is observational in nature, as it will not manipulate the treatment assignment in the MOOD clinical trial or otherwise impact concurrently ongoing treatments for any condition. Researchers collecting and analyzing EEG data will be blinded to treatment assignment when participants are in the double-blinded treatment phase of the MOOD clinical trial. EEG data will be processed and analyzed to evaluate changes in frontal alpha oscillations associated with 8 weeks of active Relivion®DP stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Meets all criteria for participation in the Neurolief-sponsored MOOD clinical trial (NCT04279522) and has been randomized to a treatment group for the double-blind phase.
* Is willing and able to participate in up to 3 additional research visits for EEG data collections.

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a primary diagnosis of MDD; ages 18-70; with current episode of primary depression lasting up to 3 years; at least moderate symptom severity reflected by score on HAMD17 scale at baseline >20; history of antidepressant medication treatment resistance or intolerance and curently on stable dose of current antidepressant medication.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-11-16 (Estimated)

PRIMARY OUTCOMES:
Change in Frontal Alpha Power | 8 weeks
  Change from Pre- to Post- Stimulation Power in Frontal Electrodes at Individual Alpha Frequency Peak (IAF), as recorded in resting state EEG. Calulated as (post-pre)/ (pre+post)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Butler Hospital/Brown University Department of Psychiatry
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No